CLINICAL TRIAL: NCT04183816
Title: Effect of Total Cold-Water Immersion Vs Ice Massage Modalities on Recovery After Exercise-induced Muscle Damage Among Adults
Brief Title: Effect of Total Cold Water Immersion Vs Ice Massage Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese German University (Other)
Responsible Party: Principal Investigator, Mohammed Ali FAKHRO, DPT, Instructor, Lebanese German University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Lebanese German University
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Exercise-induced Muscle Damage
Keywords: Total cold-water immersion; ice massage; muscle damage; delayed onset of muscle soreness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total cold-water immersion group (Experimental): Participants allocated to the TCWI group completed a session of 15-minutes in cold water with a temperature of 12°C. Each Participant was totally immersed in a pool while his/her head and neck remained above water level. The water's temperature was continuously measured by a mercury-in-glass thermometer and maintained at the aforementioned temperature by continuously adding ice blocks.
  With respect to depth of immersion, TCWI is more efficient than partial CWI since exposing a larger area of the body is needed for cardiovascular changes to occur (Murray and Cardinale, 2015; Stephens et al., 2016).
  Interventions: Other: Total cold-water immersion
- Ice massage group (Active Comparator): Participants in the IM group were seated. The investigator in charge of this intervention group applied Ice cubes massage in a clockwise circular motion on the thigh area (quadriceps) for 15 minutes.
  Interventions: Other: Ice massage

INTERVENTIONS:
Other: Total cold-water immersion — TCWI group completed a session of 15-minutes in cold water with a temperature of 12°C.
  Arms: Total cold-water immersion group
Other: Ice massage — Ice cubes massage in a clockwise circular motion on the thigh area (quadriceps) for 15 minutes.
  Arms: Ice massage group

SUMMARY:
Evidence regarding the effect of the therapeutic modalities on muscle recovery after exercise-induced muscle damage (EIMD) was lacking. Therefore, this study played a role in bridging this gap, where total cold-water immersion (TCWI) values return to baseline 72 h after the muscle damage protocol, regarding creatine kinase (CK) levels, power and strength, and delayed onset of muscle soreness (DOMS).

DETAILED DESCRIPTION:
Participants were recruited by means of convenience sampling. A message was sent via WhatsApp for all the contact list of the investigators. This message included a brief explanation of the study purpose, phone numbers of the three investigators and a request to forward this message to the contact lists of the recipients.

At the beginning of the study, all participants' data were recorded, including their physical characteristics and eligibility.

Eligible participants were given information sheets and signed consent forms. Afterward, they were familiarized with the experimental procedure and given numbers in order to assure blindness during the processes of allocating them into groups and assessing the outcomes. Final participants included 60 eligible stratified into two blocks (30 males and 30 females).

Then a randomization website -website spreadsheet generator; http://www.randomization.com was used to randomly allocate each into one of two intervention groups: 1) Total CWI (TCWI) or 2) IM.

Baseline measurements of both groups (TCWI and IM) were taken and include one repetition maximun (1-RM), (2) CMJ, (3) VAS, and (4) Serum CK tests. Testing was followed by a warm-up session and then by muscle damage protocol. Thereafter, each of the interventions (TCWI or IM) were performed and followed by post-exercise measurements at 2; 24, 48 and 72 hours.

Muscle damage protocol. Muscle damage was induced by 20 sets of 5 drop jumps each, with a two-minute rest between sets. Participants were instructed to drop jump from a 60-cm box, then perform a maximal bipodal CMJ, then land on the floor with knees flexed to at least 90°, while keeping their hands on their knees to eliminate additional force by upper limbs. This protocol produces a response similar to that obtained from high-intensity multi-joint exercises (Vieira et al., 2016).

Total cold-water immersion. The best results of recovery from EIMD were provided by TCWI with a water temperature between 11 and 15°C and an immersion time of 11 to 15 minutes according to Lee et al. (2012) and Machado et al. (2016). For that reason, participants allocated to the TCWI group completed a session of 15-minutes in cold water with temperature of 12°C.

Participants were seated while immersing their whole body in water except their head and neck. The water's temperature was continuously measured by a mercury-in-glass thermometer and was maintained at a temperature of 12°C by adding blocks of ice when needed.

With respect to depth, TCWI is more efficient than partial CWI since exposing a larger mass of the body including the core is needed for cardiovascular changes to occur, since the major heat exchange that leads to cooling occurs via conduction by surrounding water, so the higher the level of water immersion is, the greater the surface area of the body in contact with water will be, leading to better recovery effect (Murray and Cardinale, 2015; Stephens et al., 2016).

Ice massage. The IM group was seated and subjected to a circular local massage by a cube of ice for 15 minutes for each leg on the region of quadriceps muscles.

Data Analysis The results were analyzed by the Statistical Package for the Social Sciences (SPSS) version 21.0 for windows. The Shapiro-Wilk test was used to check the normality of the data distribution. A probability (p) value of >0.05 indicates that there is no significant difference between groups.

Analysis of variance (ANOVA) test was used to compute the within-group differences of each variable (muscle damage, strength, power, and DOMS) at different testing times (Baseline, 2h, 24h, 48h and 72h after exercise).

Factorial repeated measures ANOVA test was used to determine between-group difference between TCWI and IM groups, of each variable (muscle damage, strength, power, and DOMS) at different testing times (Baseline, 2h, 24h, 48h and 72h after exercise).

ELIGIBILITY:
Inclusion Criteria:

* Lebanese adults aged between 19 and 44 years,
* resided in Tyre and Saida districts, and Beirut governorate,
* regular exercise (30 min of moderate-intensity physical activity on at least 3 d. wk-1 for at least the past 3 months).

Exclusion Criteria:

* history of serious lower limb trauma (fractures, meniscus or ligament tears)
* troubles of the sensation of cold temperature,
* cardiopulmonary or inflammatory diseases
* follow regular strength and plyometric training exercises

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Change measure of Serum creatine kinase blood test | Baseline, 2 hours, 24 hours, 48 hours and 72 hours
  Muscle damage was tested by serum CK blood test, rather than the other affected intramuscular proteins, due to its dramatic increase in blood plasma after EIMD, and the low cost of its assay (Clarkson & Hubal, 2002).
  The blood samples were taken to a specific laboratory test where it was allowed 30 min for clotting, then centrifuged for 20min at room temperature. The serum was then stored at -20°C until analysis. Finally, Serum CK activity was analyzed with an enzymatic method at 37°C (Vieira et al., 2016).
Change measure of Countermovement jump test | Baseline, 2 hours, 24 hours, 48 hours and 72 hours
  The countermovement jump (CMJ) test is used to measure muscle power. CMJ is a vertical jump that begins with a countermovement, defined as flexion of the knees (Thomas K, French D, Hayes P.R, 2009). CMJ was shown to affect vertical jump height which indicates that adaptations relating to increases in leg power have occurred. The end of the landing phase represents the end of the CMJ and is defined when the pelvis, marked by the four superior iliac spines, achieved its lowest position (Schwartz et al, 2017).
  Participants were asked to flex their knees, and then to perform a maximally explosive vertical jump upward, and then land on the floor. To ensure measurement accuracy and reliability, participants were instructed to keep their legs and hips extended until contact is made (end of landing phase) and to keep their hands on their hips during the jump (Markovic, 2004). They repeated the CMJ three times and the highest jump was recorded.
Change measure of 1-Repetition Maximum test | Baseline, 2 hours, 24 hours, 48 hours and 72 hours
  Muscle strength is measured by one 1-RM, which is considered the gold standard for measuring strength (Puthoff, 2006).
  Before testing, the participants performed a general cardiovascular warm-up (jogging) for five minutes (Chen, Chen & Jan, 2015).
  The participants were asked to perform knee extension for the dominant leg to test the quadriceps muscle starting from 90-degrees knee flexion, with a rest time of one minute. Then, weighs are gradually adjusted, starting from 10 warm-up repetitions, with a light load (LeBrasseur et al., 2008); followed by a sequence of progressively increased weight loads until the subject fails to safely and correctly complete a full range of motion. This load is recorded and referred to as the 1-RM (Puthoff, 2006).
Change measure of Visual Analogue Scale | Baseline, 2 hours, 24 hours, 48 hours and 72 hours
  Participants were asked to perform maximal isometric contraction of their right knee extensors muscles for 4 seconds and immediately rate their soreness according to the visual analogue scale (VAS) of 10 degrees, ranging from "no soreness" (0) to "severe soreness" (10) (Vieira et al., 2016). VAS showed excellent reliability in the assessment of DOMS, the ICC range was 0.98-0.99 for VAS (Lau, Muthalib & Nosaka, 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese German University, Jounieh, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fakhro MA, AlAmeen F, Fayad R. Comparison of total cold-water immersion's effects to ice massage on recovery from exercise-induced muscle damage. J Exp Orthop. 2022 Jun 22;9(1):59. doi: 10.1186/s40634-022-00497-5. PMID 35731373

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT04183816/Prot_SAP_000.pdf